CLINICAL TRIAL: NCT00053495
Title: The Effect of Dose On Safety, Tolerability, and Immunogenicity of ACAM2000 Smallpox Vaccine in Adults Without Previous Smallpox Vaccination
Brief Title: Effect of Dose, Safety, Tolerability of a New Smallpox Vaccine in Adults Without Previous Smallpox Vaccination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-400-005
Record Dates: First submitted 2003-01-30; First posted 2003-01-31 (Estimated); Results first posted 2011-02-11 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Smallpox
Keywords: Smallpox
MeSH Terms: conditions — Smallpox | interventions — Smallpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1: ACAM2000 Dose 1 (Experimental): Participants will receive a single dose of ACAM2000 smallpox vaccine, 1.0x10-8th plaque-forming units (PFU)/mL on Day 0.
  Interventions: Biological: Vaccinia virus: ACAM2000 smallpox vaccine
- Group 2: ACAM2000 Dose 2 (Experimental): Participants will receive a single dose of ACAM2000 smallpox vaccine, 2.0x10-8th plaque-forming units/mL on Day 0.
  Interventions: Biological: Vaccinia virus: ACAM2000 smallpox vaccine
- Group 3: ACAM2000 Dose 3 (Experimental): Participants will receive a single dose of ACAM2000 smallpox vaccine, 1.0x10-7th plaque-forming units/mL on Day 0
  Interventions: Biological: Vaccinia virus: ACAM2000 smallpox vaccine
- Group 4: ACAM2000 Dose 4 (Experimental): Participants received a single dose of ACAM2000 smallpox vaccine, 5.0x10-6th plaque-forming units/mL on Day 0
  Interventions: Biological: Vaccinia virus: ACAM2000 smallpox vaccine
- Group 5: Dryvax® Vaccine (Active Comparator): Participants will receive a single dose of Dryvax® smallpox vaccine, 1.0x10-8th plaque-forming units/mL on Day 0
  Interventions: Biological: vaccinia virus (calf lymph): Dryvax

INTERVENTIONS:
Biological: Vaccinia virus: ACAM2000 smallpox vaccine — Group 1 dose: 1.0x10-8th PFU/ml Group 2 dose: 2.0x10-8th PFU/ml Group 3 dose: 1.0x10-7th PFU/ml Group 4 dose: 5.0x10-6th PFU/ml
  Arms: Group 1: ACAM2000 Dose 1; Group 2: ACAM2000 Dose 2; Group 3: ACAM2000 Dose 3; Group 4: ACAM2000 Dose 4
Biological: vaccinia virus (calf lymph): Dryvax — Group 5 dose: 1.0x10-8th PFU/ml
  Other Names: Dryvax®
  Arms: Group 5: Dryvax® Vaccine

SUMMARY:
The purpose of this study is to examine the safety and the effectiveness of a new vaccine for the prevention of the disease, smallpox.

DETAILED DESCRIPTION:
The objective of this study is to determine the minimum dose of ACAM2000 that is calculated to produce a major cutaneous reaction in at least 90% of a population of healthy adults 18-29 years of age and naïve to smallpox vaccine. Specifically, the objectives of this study are to:

1. Compare the safety and tolerability of four dose levels of ACAM2000 and a standard dose of Dryvax® in healthy adults 18-29 years of age and naïve to smallpox vaccine. Safety and tolerability will be determined by examination of the local cutaneous reaction, adverse events, physical examinations, vital signs, structured interviews, and laboratory analysis.
2. Determine the immunogenicity of four dose levels of ACAM2000 and a standard dose of Dryvax® in healthy adults 18-29 years of age by comparing:

   1. the proportion of subjects at each dose level who develop a major cutaneous reaction;
   2. the proportion of subjects in each treatment group who develop neutralizing antibodies, including the fold-increase in antibody titer between Baseline and Day 30 sera; and the geometric mean vaccinia neutralizing antibody titer on Day 30.
3. Determine the minimum dose of ACAM2000 that is calculated to produce a major cutaneous reaction in at least 90% of a population of healthy adults 18-29 years of age and naïve to smallpox vaccine.

ELIGIBILITY:
Inclusion criteria:

* females must not be pregnant, lactating and must agree to use an effective form of birth control for the 30 days following vaccination or unable to bear children.
* agree to be available for the entire study and agree to comply with all requirements.

Exclusion criteria:

* military service prior to 1989.
* history of previous smallpox vaccination.
* children 1 year of age or younger in the household or be in close contact
* smallpox vaccination within ten years
* known or suspected human immunodeficiency virus (HIV) infection, primary immunodeficiency disorder, leukemia, lymphoma, or current radiation treatment or use of immunosuppressive or anti-neoplastic drugs or have a household member or intimate contact with the conditions listed above.
* renal disease
* current or past history of eczema or a household member or direct contact who has eczema.
* known allergy or past allergic reactions to latex gloves or to antibiotics which include neomycin, streptomycin, chlortetracycline, and polymyxin B
* known allergy or past allergic reaction to blood products.
* known allergy to cidofovir or sulfa-containing drugs.
* history of allergic phenomena following smallpox vaccination in the past, including urticaria, erythema multiforme, or Stevens-Johnson syndrome.
* transfusion of blood or treatment with any blood product.
* current or history of drug or alcohol abuse
* inoculation with any other live vaccine or participating in another drug or vaccine trial within 30 days of enrollment.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 353 (Actual)
Dates: Start 2003-01; Primary Completion 2003-06 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Emergent BioSolutions
Locations (4):
- United States (4):
  - Orlando Clinical Research Center, Orlando, Florida
  - PRA International, Lenexa, Kansas
  - Bio-Kinetic Clinical Applications, Springfield, Missouri
  - Memorial Hospital of Rhode IslandDivision of Infectious Diseases, Pawtucket, Rhode Island

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 10 January 2003 to 14 April 2003 in 4 medical centers in the US.
Pre-assignment Details: A total of 353 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- ACAM2000 Dose 1: Participants received a single dose of ACAM2000 smallpox vaccine, 1.0x10^8th plaque-forming units/mL on Day 0
- ACAM2000 Dose 2: Participants received a single dose of ACAM2000 smallpox vaccine, 2.0x10^8th plaque-forming units/mL on Day 0
- ACAM2000 Dose 3: Participants received a single dose of ACAM2000 smallpox vaccine, 1.0x10^7th plaque-forming units/mL on Day 0
- ACAM2000 Dose 4: Participants received a single dose of ACAM2000 smallpox vaccine, 5.0x10^6th plaque-forming units/mL on Day 0
- Dryvax® Vaccine: Participants received a single dose of Dryvax® smallpox vaccine, 1.0x10^8th plaque-forming units/mL on Day 0
Period: Overall Study
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Started | 51 | 101 | 101 | 51 | 49
Completed | 51 | 101 | 101 | 51 | 49
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine | Total
Number analyzed (Participants) | 51 | 101 | 101 | 51 | 49 | 353
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 51 | 101 | 101 | 51 | 49 | 353
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23 (2.4) | 22 (3.1) | 22 (3.2) | 22 (3.0) | 22 (3.1) | 22 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 36 | 34 | 14 | 13 | 115
  Male | 33 | 65 | 67 | 37 | 36 | 238
Region of Enrollment [Number; unit: participants]
  United States | 51 | 101 | 101 | 51 | 49 | 353

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Adverse Events of Severe Intensity Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine
Description: The severity of each reported adverse event was classified by the investigator according to the following definitions. None - no symptom; Mild - awareness of sign or symptoms, but easily tolerated; Moderate - discomfort enough to cause interference with usual activity; and Severe - incapacitating with inability to work or perform usual activity.
Time Frame: Days 0 to 30 post-vaccination
Population: Adverse events were assessed in the safety, intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 101 | 101 | 51 | 49
Participants
  Lymph Node Pain | 2 | 4 | 3 | 4 | 2
  Lymphadenopathy | 0 | 0 | 0 | 1 | 0
  Diarrhea Not Otherwise Specified | 1 | 0 | 0 | 0 | 0
  Nausea | 1 | 0 | 0 | 0 | 0
  Vomiting Not Otherwise Specified | 1 | 0 | 0 | 0 | 0
  Injection Site Erythema | 1 | 6 | 14 | 11 | 15
  Injection Site Swelling | 0 | 0 | 1 | 1 | 0
  Injection Site Pruritus | 0 | 0 | 1 | 0 | 1
  Fatigue | 0 | 0 | 1 | 0 | 0
  Injection Site Pain | 0 | 0 | 1 | 0 | 0
  Dehydration | 0 | 0 | 1 | 0 | 0
  Myalgia | 0 | 0 | 0 | 1 | 0
  Headache Not Otherwise Specified | 1 | 0 | 4 | 1 | 0
  Pregnancy Not Otherwise Specified | 0 | 1 | 0 | 1 | 0
  Dysuria | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Neutralizing Antibody Response Titers Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine.
Time Frame: Day 30 post-vaccination
Population: Neutralizing antibody response titers were evaluated in the antibody evaluable, per-protocol population.
Measure: Mean (Standard Deviation); unit: PRNT50 Titers
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 100 | 100 | 50 | 49
PRNT50 Titers | 212 (536.4) | 278 (581.6) | 425 (947.4) | 582 (1129.3) | 1515 (6019.4)

3. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Rash Events Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine.
Time Frame: Days 0 to 30 post-vaccination
Population: Treatment-emergent rash events were assessed in the safety, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 101 | 101 | 51 | 49
Participants
  Rash Not Otherwise Specified | 3 | 10 | 9 | 5 | 7
  Rash Pruritic | 0 | 1 | 0 | 0 | 0
  Rash Pustular | 0 | 1 | 0 | 0 | 1
  Application Site Rash | 0 | 1 | 1 | 3 | 2
  Injection Site Rash | 0 | 0 | 1 | 0 | 1
  Any Rash Event | 3 | 11 | 10 | 7 | 10

4. Other Pre Specified Outcome: Clinical Chemistry Parameters (Aspartate Aminotransaminase and Alanine Aminotransferase) at Baseline and Day 15 Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine
Time Frame: Days 0 (baseline) and 15 post-vaccination
Population: Clinical chemistry parameters were assessed in safety, intent-to-treat population
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 101 | 101 | 51 | 49
IU/L
  Aspartate Aminotransferase (Baseline) | 21 (7.4) | 21 (5.9) | 22 (7.1) | 23 (7.1) | 20 (5.8)
  Aspartate Aminotransferase (Day 15) | 23 (10.5) | 21 (7.7) | 22 (7.5) | 21 (6.3) | 22 (6.8)
  Alanine Aminotransferase (Baseline) | 32 (15.0) | 32 (16.2) | 33 (17.4) | 36 (18.5) | 31 (16.8)
  Alanine Aminotransferase (Day 15) | 33 (15.4) | 32 (17.5) | 33 (16.6) | 34 (16.2) | 33 (17.9)

5. Other Pre Specified Outcome: Clinical Chemistry Parameters (Creatinine and Glucose) at Baseline and Day 15 Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine
Time Frame: Days 0 (baseline) and 15 post-vaccination
Population: Clinical chemistry parameters were assessed in safety, intent-to-treat population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 101 | 101 | 51 | 49
mg/dL
  Creatinine (Baseline) | 0.97 (0.147) | 0.96 (0.153) | 0.98 (0.181) | 0.97 (0.171) | 0.97 (0.158)
  Creatinine (Day 15) | 0.98 (0.149) | 0.98 (0.142) | 0.98 (0.169) | 1.00 (0.144) | 1.00 (0.163)
  Glucose (Baseline) | 85 (7.3) | 84 (9.8) | 86 (7.4) | 86 (8.3) | 87 (18.6)
  Glucose (Day 15) | 83 (14.2) | 86 (14.6) | 86 (10.6) | 87 (13.2) | 88 (21.4)

6. Primary Outcome: Participants With ≥ 4-fold Increase in Plaque-Reduction Neutralization Test (PRNT50) Titers Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine.
Time Frame: Day 30 post-vaccination
Population: Plaque-reduction neutralization test (PRNT50) titers were determined in the antibody evaluable, per-protocol population
Measure: Number; unit: Participants
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 50 | 100 | 100 | 51 | 49
Participants | 28 | 73 | 84 | 48 | 47

7. Other Pre Specified Outcome: Selected Hematology Parameters (Hematocrit, Lymphocyte, and Eosinophil) at Baseline and on Day 15 in Participants Vaccinated With ACAM2000 or Dryvax® Smallpox Vaccine.
Time Frame: Days 0 (baseline) and 15 post-vaccination
Population: Hematology parameters were evaluated in the safety, intent-to-treat population.
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 101 | 101 | 51 | 49
Percentage (%)
  Hematocrit (Baseline) | 43.7 (4.20) | 43.2 (3.71) | 43.2 (4.44) | 44.2 (3.29) | 44.1 (3.54)
  Hematocrit (Day 15) | 42.8 (3.74) | 42.3 (3.59) | 42.7 (3.21) | 43.2 (2.55) | 43.1 (3.13)
  Lymphocytes (Baseline) | 30.6 (8.26) | 31.5 (8.33) | 30.7 (7.00) | 29.6 (7.45) | 31.6 (7.99)
  Lymphocytes (Day 15) | 33.9 (8.62) | 34.0 (7.41) | 34.7 (7.93) | 33.9 (6.83) | 33.8 (7.58)
  Eosinophils (Baseline) | 2.5 (1.61) | 2.5 (1.95) | 2.4 (1.69) | 2.3 (1.42) | 2.4 (1.72)
  Eosinophils (Day 15) | 2.8 (2.07) | 2.8 (2.11) | 2.6 (1.65) | 2.7 (1.42) | 2.7 (1.61)

8. Other Pre Specified Outcome: Selected Hematology Parameters (Red Blood Count and Platelets) at Baseline and on Day 15 in Participants Vaccinated With ACAM2000 or Dryvax® Smallpox Vaccine.
Time Frame: Days 0 (baseline) and 15 post-vaccination
Population: Hematology parameters were evaluated in the safety, intent-to-treat population.
Measure: Mean (Standard Deviation); unit: x10-6th/μL
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 101 | 101 | 51 | 49
x10-6th/μL
  Red Blood Cell Count (Baseline) | 5.1 (0.53) | 5.0 (0.47) | 5.1 (0.44) | 5.1 (0.45) | 5.1 (0.44)
  Red Blood Cell Count (Day 15) | 5.0 (0.50) | 4.9 (0.44) | 5.0 (0.39) | 5.0 (0.37) | 5.0 (0.38)
  Platelets (Baseline) | 274 (64.0) | 282 (60.1) | 281 (68.1) | 274 (52.4) | 267 (51.6)
  Platelets (Day 15) | 284 (58.6) | 280 (57.7) | 281 (65.1) | 284 (59.3) | 285 (52.1)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for up to 6 months post-vaccination.
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Serious Adverse Events (participants affected / at risk) | 1/51 | 1/101 | 0/101 | 1/51 | 0/49
Other Adverse Events (participants affected / at risk) | 51/51 | 99/101 | 98/101 | 51/51 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACAM2000 Dose 1 (N=51) | ACAM2000 Dose 2 (N=101) | ACAM2000 Dose 3 (N=101) | ACAM2000 Dose 4 (N=51) | Dryvax® Vaccine (N=49)
Pregnancy Not Otherwise Specified (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACAM2000 Dose 1 (N=51) | ACAM2000 Dose 2 (N=101) | ACAM2000 Dose 3 (N=101) | ACAM2000 Dose 4 (N=51) | Dryvax® Vaccine (N=49)
Lymph Node Pain (Blood and lymphatic system disorders) | 22 | 59 | 61 | 39 | 44
Lymphadenopathy (Blood and lymphatic system disorders) | 11 | 26 | 25 | 19 | 17
Nausea (Gastrointestinal disorders) | 13 | 21 | 21 | 11 | 14
Diarrhea Not Otherwise Specified (Gastrointestinal disorders) | 9 | 13 | 21 | 5 | 7
Vomiting Not Otherwise Specified (Gastrointestinal disorders) | 5 | 2 | 10 | 4 | 3
Injection Site Pruritus (General disorders) | 43 | 89 | 82 | 51 | 49
Injection Site Erythema (General disorders) | 27 | 65 | 64 | 37 | 37
Injection Site Pain (General disorders) | 22 | 59 | 58 | 35 | 35
Fatigue (General disorders) | 23 | 41 | 55 | 29 | 28
Malaise (General disorders) | 18 | 27 | 29 | 18 | 23
Feeling Hot (General disorders) | 14 | 26 | 24 | 13 | 19
Rigors (General disorders) | 7 | 14 | 19 | 13 | 14
Injection Site Swelling (General disorders) | 3 | 6 | 6 | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 40 | 47 | 26 | 27
Headache Not Otherwise Specified (Nervous system disorders) | 30 | 51 | 49 | 24 | 28
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 11 | 8 | 2 | 1
Rash Not Otherwise Specified (Skin and subcutaneous tissue disorders) | 3 | 10 | 9 | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.